CLINICAL TRIAL: NCT05551260
Title: Assessing Moral Cognitive Skills in Adults With Autism Spectrum Disorders
Acronym: CoMorA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-A01040-43
Record Dates: First submitted 2022-07-19; First posted 2022-09-22 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Moral cognition; autism spectrum disorders
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: This study uses standard neuropsychological tests and a computerized experimental task, submitted to two parallel groups: participants with ASD and control participants matched in age, gender and level of education (1:1 ratio). Participants in both groups completed the neuropsychological tests and the experimental task successively (fixed order for all participants). Within the experimental task, the experimental conditions appear randomly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- People with ASD (Experimental): 30 people with ASD without IDD
  Interventions: Other: Neuropsychological assessments (tests allowing to measures attentional, executive and emotional performances) and experimental protocol assessing moral cognition
- Neurotypicals (Active Comparator): 30 neurotypicals
  Interventions: Other: Neuropsychological assessments (tests allowing to measures attentional, executive and emotional performances) and experimental protocol assessing moral cognition

INTERVENTIONS:
Other: Neuropsychological assessments (tests allowing to measures attentional, executive and emotional performances) and experimental protocol assessing moral cognition — Day 0: sending of the information notice
  Day 1 : signing the consent form + neuropsychological tests assessing reasoning and abstraction abilities, attentional processes, executive functions (including inhibition and mental flexibility) and social cognitive functions, including facial emotion recognition, theory of mind and perception and social knowledge (duration 1h30-2h). Experimental protocol: vignettes of moral offenses manipulating variables of intention and consequence. This systematic manipulation, commonly used in the field of moral judgment, usually leads to 3 combinations of variables: intentional harm (present intention; present consequence); attempted harm (intent present; consequence absent); accidental harm (intention absent; consequence present). Another form of accidental harm will also be constructed (positive intention; present consequence) (duration : 1h)
  Between day 1 and day 21 : second part of the Day 1 tests

SUMMARY:
In the international literature, it is currently accepted that, relative to neurotypicals, people with Autism Spectrum Disorder (ASD) present patterns of moral judgments marked by a minimization of intentionality and a strong condemnation of agents responsible for accidents. However, until now, all studies are based on declarative paradigms, and no one has proposed to examine the relationship of people with ASD to moral transgressions (i.e. to a bad action done deliberately or to a good deed deliberately omitted) in an implicit paradigm, that is, when the answer is made on the assignment of an expressive face to these moral offenses. Furthermore, no study has investigated whether diminished sensitivity to intention and intransigence of incidental judgment occur in both automatic (implicit) and deliberative (explicit) settings.

Investigators planned to study how people with ASD without intellectual disability process emotions expressed by others in response to different forms of moral offense and to examine whether patterns potentially contrast in degree and/or kind with those of neurotypicals.

DETAILED DESCRIPTION:
In the CoMorA project, participants will participate to two independent tasks: an explicit one of deciding whether or not an emotion expressed on the face of a third person would be an appropriate emotional reaction to the offense, and an implicit one in which the subjects will have to determine the fastest sex to which the face expressing such or such an emotion belongs. This procedure initiates an implicit processing of the facial expression.

The theoretical hypotheses of the CoMorA project are the following:

* In the explicit response condition, people with ASD will show different emotional assignment patterns than controls do, depending on the nature of the offense (accidental transgression, attempted harm, and intentional harm).
* In the implicit response condition, people with ASD will exhibit emotion processing patterns identical to those of controls.
* The differences in responses of controls and people with ASD in the explicit condition will be underpinned by executive functions and social cognitive performances.

ELIGIBILITY:
Inclusion Criteria:

ASD group:

* Diagnosis of ASD according to DSM-5 criteria
* Age between 18 and 40 years old
* Francophone
* Affiliated to social security
* Having given their consent to participate in the study
* Patient under guardianship and curatorship

Neurotypical group:

* Age between 18 and 40 years old
* Francophone
* Affiliated to a social security scheme
* Having given their consent to participate in the study

Exclusion Criteria:

ASD group:

* Diagnosis of intellectual development disorder established according to DSM-5 criteria
* Language, sensory or motor impairments hindering participation in the study

Control group:

* Neurodevelopmental pathology (declarative)
* Neurological pathology
* Language, sensory or motor impairments hindering participation in the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of moral cognition | at day 0
  First the reading of a vignette presenting a moral scenario jointly manipulating variables of intention and consequence. This systematic manipulation, commonly used in the field of moral judgment, leads to 4 combinations of variables:
  intentional harm: present intention; present consequence attempted harm: present intention; absent consequence accidental harm: absent intention; present consequence accidental harm with positive intention: positive intention; present consequence
  A presentation to the participants of a face presenting an intense facial expression (in a counterbalanced way of man or woman.
  Explicit procedure: After the implicit classification task, the participants will see the same photo and will have to indicate whether the expression of this person is appropriate to the situation described. The proportion of correct answers (CP) will be recorded.
Evaluation of moral cognition | between day 1 and day 21
  First the reading of a vignette presenting a moral scenario jointly manipulating variables of intention and consequence. This systematic manipulation, commonly used in the field of moral judgment, leads to 4 combinations of variables:
  intentional harm: present intention; present consequence attempted harm: present intention; absent consequence accidental harm: absent intention; present consequence accidental harm with positive intention: positive intention; present consequence
  A presentation to the participants of a face presenting an intense facial expression (in a counterbalanced way of man or woman
  1. Implicit procedure: The participants will participate to an implicit task consisting in classifying as quickly as possible the sex to which the character of the photograph belongs (male or female). The response time (TR) will be recorded.

SECONDARY OUTCOMES:
Reasoning and general intellectual level | at day 0 and between day 1 and day 21
  the following neuropsychological tests will be proposed: Similarities: Weschler Adult Intelligence Scale (WAIS-IV ) During this test, the subject must determine the common point or the similarity between two concepts (i.e., orange-banana). This test measures the ability to form abstract concepts. Score vary from 1 to 19 Cubes: WAIS-IV Using 2, 4 or 9 two-coloured cubes, the subject must reproduce the shapes presented to him, respecting the organization of the figure. This test measures non-verbal reasoning, visual-perceptive, visual-constructive and practical skills. Score vary from 1 to 19 Matrices: WAIS-IV The subject must complete a matrix made up of elements according to a logic. This test assesses non-verbal reasoning as well as visual-spatial abilities. Score vary from 1 to 19 Vocabulary: WAIS-IV The subject must explain the meaning of certain words by giving their definition. This test assesses the level of vocabulary and the integrity of the lexical stock. From 1 to 19
Attentional and executive measures | at day 0 and between day 1 and day 21
  Test d'Attention Concentrée (D2R) : consists of the letters "d" and "p" provided with dashes.Scores vary from 1 to 99. Stroop: name the color of colored rectangles, read color names printed in black,and name the color of the ink in which the color words are written and inhibit the reading of each word. It measures inhibition. Trail Making Test (TMT) is carried out in 2 stages. During the part A the subject must connect numbers in ascending order with a pencil. Then, during the part B the subject must alternately connect a number to a letter in an increasing way. It makes it possible to measure reactive flexibility capacities. Digit span : (WAIS-IV) consists of repeating orally a sequence of numbers given orally and measures the storage capacity of short-term information (short-term memory). From 1 to 19. Backwards digit span (WAIS-IV) Same but in reverse order (e.g., 5-7-9 > 9-7-5). This test measures the ability to manipulate short-term information (working memory). From 1 to 19.
Social cognitive measures | at day 0 and between day 1 and day 21
  TREF (Facial Emotion Recognition Test) assesses the ability to recognize facial emotions. It provides an overall emotion recognition score and a sub-score per emotion, as well as their detection threshold. Scores vary from 0 to 100% PerSo (ClaCoS) is to assess the perception and processing of social cues present in a situation in order to make inferences about it. It is made up of 4 color plates selected according to the type of emotion and situation represented (simple/complex context; simple/complex emotion). The task to be performed is inspired by the IPT cognitive remediation program. Scores vary from 0 to 24.
  RMET (Reading the Mind in the Eyes Test) is made up of 36 photos of looks in black and white. The subject must choose, among 4 propositions, the one which seems the most adapted to describe the mental state of the character. This task is classically used to assess affective theory of mind abilities in autism. Score vary from 0 to 36.
Alexithymia | at day 0 and between day 1 and day 21
  TAS-20 (Toronto Alexithymia Scale 20 items) is composed of 20 items evaluating 3 dimensions of alexithymia:
  * Difficulty describing emotions - Ex: "It is difficult for me to find the right words to describe my feelings"
  * Difficulty identifying emotions - Ex: "I sometimes do not know what emotion I am feeling exactly"
  * Operative thinking - Ex: "I prefer to talk to people about their activity rather than their feel
  For the questionnaire the raw scores will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Elodie PEYROUX, Principal Investigator — Centre Hospitalier le Vinatier
Locations (1):
- centre de réhabilitation - Hôpital le Vinatier, Lyon, Rhône, France

IPD SHARING:
Plan to Share IPD: No